CLINICAL TRIAL: NCT01314625
Title: A Pilot Study Evaluating Hypotension and Autonomic Nervous System Dysfunction After Therapy With Bortezomib-containing Regimens in Subjects With Multiple Myeloma
Brief Title: A Study Evaluating Hypotension and Autonomic Nervous System Dysfunction in Multiple Myeloma (MM) Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Other Study IDs: UAMS 2009-50
Record Dates: First submitted 2011-03-10; First posted 2011-03-14 (Estimated); Last update posted 2012-05-16 (Estimated); Status verified 2012-05

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- one arm

SUMMARY:
The purpose of this study is to determine whether the orthostatic hypotension reported among subjects during bortezomib-containing regimen is caused by a dysfunction of the autonomic nervous system (ANS).

DETAILED DESCRIPTION:
1. To gather pilot data on the incidence of autonomic dysfunction in patients with Multiple Myeloma prior to treatment with Bortezomib.
2. To characterize the changes in the ANS including the fluctuations in blood pressure (hypotension /hypertension) associated with bortezomib.
3. To determine the duration of the ANS dysfunction if present.

This is not a treatment study, only an evaluation of the autonomic nervous system (ANS) among subjects receiving antimyeloma therapy which includes bortezomib (Velcade).

ELIGIBILITY:
Inclusion Criteria:

* Subjects with Active Multiple Myeloma who are scheduled to be treated with Bortezomib-containing regimens.
* Subjects must have signed an IRB-approved informed consent indicating their understanding of the proposed treatment and understanding that the protocol has been approved by the IRB.

Exclusion Criteria:

* Subjects with unstable cardiovascular disease. Recent (< 6 months) myocardial infarction, unstable angina, difficult to control congestive heart failure, uncontrolled hypertension, or difficult to control cardiac arrhythmias.
* Subjects unable to perform the Valsalva maneuver such as patients with clinically significant aortic stenosis, glaucoma or retinopathy.
* Subjects receiving Selective Serotonin Reuptake Inhibitors.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: To determine whether the orthostatic hypotension reported among subjects during bortezomib-containing regimen is caused by a dysfunction of the autonomic nervous system (ANS).
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2011-03; Primary Completion 2012-06 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
To determine whether the orthostatic hypotension reported among subjects during bortezomib-containing regimen is caused by a dysfunction of the autonomic nervous system (ANS). | 1 year
  Patient symptoms that are most disabling after Bortezomib treatment appear to be those caused by autonomic instability/dysfunction such as orthostatic intolerance, vasomotor changes with pallor, sweating, gut hypermotility and sensory peripheral neuropathy. Although these symptoms are not specific, clinical wisdom dictates that the autonomic nervous system (ANS) be investigated first.
  However, the mechanism (s) underlying the orthostatic hypotension and other Velcade-associated toxicities remain unclear.
  We plan to evaluate the exact cause behind these severe adverse events.

SECONDARY OUTCOMES:
To gather pilot data on the incidence of autonomic dysfunction in patients with Multiple Myeloma prior to treatment with Bortezomib. | 1 year
  Bortezomib (Velcade), a particularly effective agent against multiple myeloma, is associated with a 13 % incidence of hypotension.
  A recent analysis of over 170 subjects enrolled in UAMS protocol for therapy of newly diagnosed myeloma focused on three Velcade-containing cycles (two induction cycles and one consolidation with VDT-PACE (V=Velcade). A 9-19 % incidence of hypotension was observed. In addition, these cycles were complicated by diarrhea and sensory dysesthesias.
  We plan to calculate the incidence of Hypotension in these pt's treated with Bortezomib
To characterize the changes in the ANS including the fluctuations in blood pressure (hypotension /hypertension) associated with bortezomib. | 1 year
  Although orthostatic blood pressure (BP) measurements were not routinely obtained in our study, analysis of daily BP values during Velcade-containing cycles revealed that > 60% of subjects exhibited BP lability with variations in their BP measurements by >20mm systolic and >10mm diastolic on successive days during the course of therapy. A subset of these subjects presented with severe symptoms, particularly orthostatic hypotension, and at times requiring hospitalization.
  We plan to investigate the ANS changes with a serial orthostatic measurement after Bortezomib therapy

CONTACTS AND LOCATIONS:
Overall Officials: Elias Anaissie, MD, Principal Investigator — Principal Investigator
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States